CLINICAL TRIAL: NCT00200070
Title: STARTSTIM - Stimulation Therapy for Angina Refractory To Standard Treatments, Interventions and Medications
Brief Title: Neurostimulation to Treat Refractory Angina Pectoris Pain
Acronym: STARTSTIM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Medtronic Neuromodulation, Medtronic Neuromodulation
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1659
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Angina Pectoris
Keywords: Angina Pectoris Pain
MeSH Terms: conditions — Angina Pectoris | interventions — Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation

SUMMARY:
The therapy under investigation involves an implanted Medtronic neurostimulation system to relieve symptoms of angina pectoris pain. Electrical impulses are applied to targeted areas of the spinal cord through an implanted lead (a flexible insulated wire) that is powered by an implanted battery.

ELIGIBILITY:
Inclusion Criteria:

* stable angina pectoris associated with reversible myocardial ischemia and significant coronary artery disease (CAD)
* classified as Canadian Cardiovascular Society (CCS) angina class III or IV
* refractory angina despite receiving optimal/maximal medical treatment
* not a candidate for bypass surgery, angioplasty or stent

Exclusion Criteria:

* not able to perform exercise treadmill testing
* previously received therapeutic transcutaneous electrical nerve stimulation (TENS) (within 2 years) or any spinal cord stimulation (SCS)
* has an implanted pacemaker/defibrillator (ICD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228
Dates: Start 2002-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is total exercise time on a treadmill compared between treatment groups at six months.

SECONDARY OUTCOMES:
Secondary outcome measures include exercise time to angina onset and improvement in angina symptoms and cardiovascular function.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Zipes, Principal Investigator — Indiana University School of Medicine; Nelson Svorkidal, Principal Investigator — Health Science Center, Winnipeg CANADA
Locations (8):
- United States (6):
  - Contact Medtronic for Exact Location, Gainesville, Florida
  - Contact Medtronic for Exact Location, Indianapolis, Indiana
  - Contact Medtronic for Exact Location, Boston, Massachusetts
  - Contact Medtronic for Exact Location, Minneapolis, Minnesota
  - Contact Medtronic for Exact Location, Rochester, Minnesota
  - Contact Medtronic for Exact Location, Charleston, South Carolina
- Canada (2):
  - Contact Medtronic for Exact Location, Winnipeg, Manitoba
  - Contact Medtronic for Exact Location, Ottawa, Ontario

REFERENCES:
- [Derived] Zipes DP, Svorkdal N, Berman D, Boortz-Marx R, Henry T, Lerman A, Ross E, Turner M, Irwin C. Spinal cord stimulation therapy for patients with refractory angina who are not candidates for revascularization. Neuromodulation. 2012 Nov-Dec;15(6):550-8; discussion 558-9. doi: 10.1111/j.1525-1403.2012.00452.x. Epub 2012 Apr 11. PMID 22494013